CLINICAL TRIAL: NCT04982978
Title: The Effectiveness of the Protection Motivation Theory in Reducing Vaping Behaviour in a Student Population
Brief Title: Information Interventions to Reduce Vaping in a Student Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University (Other)
Responsible Party: Principal Investigator, Harry Prapavessis, PhD, Principal Investigator, Western University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 116734
Record Dates: First submitted 2021-06-23; First posted 2021-07-29 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Vaping Related Disorder
Keywords: Protection Motivation Theory; Threat Appraisal; Health Psychology; Intention; Behaviour
MeSH Terms: conditions — Behavior | interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into one of two blocks (A or B), each containing a maximum of 75 participants (PMT present intervention group or the control group). The PMT present group will include an 8-minute informational video that explains the current research and health risks associated with vaping, within the context of a threat appraisal focus (Perceived Vulnerability and Perceived Severity). The PMT absent group (control group) will feature an 8-minute nutrition and lifestyle information video as an attention control strategy in this study. During this video intervention, the general risks and benefits of nutrition and lifestyle choices will be presented.
Who Masked: Participant
Masking Description: Participants will be allocated to one of two experimental groups using a blocked randomization method; participants will be randomized within blocks such that an equal number are assigned to each treatment. Once participants are allocated to one block, each participant will then be assigned an ID number that will represent their block as well as their individual participant ID number (i.e., Participant '100-123' would be in the same group as participant '100-124'). At Day 7 (T1), participants in each group will be emailed their respective intervention video links. Participants will not be given any information regarding group allocation or additional intervention information until the Letter of Study End notification is sent out to private email accounts of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PMT Threat Appraisal (Active Comparator): The PMT present group will include an 8-minute informational video that explains the current research and health risks associated with vaping, within the context of a threat appraisal focus (Perceived Vulnerability and Perceived Severity). During this video intervention, the severity and vulnerability of vaping among young adults, both in the short and long-term health effects will be presented. In addition, the video will explain the negative impact of vaping and focus the attention of the participants on the lack of research and information that currently exists on popular vaping products and the potentially devastating impact it can have on the health of young adult populations.
  Interventions: Behavioral: PMT Threat Appraisal
- Nutrition and Lifestyle Control (Sham Comparator): The PMT absent group will feature an 8-minute nutritional information video as an attention control strategy titled, "Vaping Health Effects". During this video intervention, the general risks and benefits of nutrition and lifestyle will be presented. The focus of this video will be on how a balanced diet and proper lifestyle choices (i.e., adequate sleep, diet, etc.) can benefit the participants lives in the short-term and long-term.
  Interventions: Behavioral: General Nutrition and Lifestyle

INTERVENTIONS:
Behavioral: PMT Threat Appraisal — The first half of the PMT present video will include narration by "Science Insider" producer, Benji Jones, including dialogue regarding the risks associated with vaping by Chief Pediatric Pulmonology at the NYU Winthrop Hospital, Dr. Melodi Pirzada, and information on nicotine by the Director of Pediatric Pulmonology at NYU's Langone Hassenfeld Children's Hospital, Dr. Mikhail Kazachkov. The second half of the PMT present video will include personal experiences and narratives by students at the University of Utah with information regarding our current knowledge of vaping health effects through research by Dr. Sean Maddock and Dr. Sean Callahan from the University of Utah to highlight the susceptibility of vaping for a population of young adults in university.
  Other Names: Threat Appraisal; Health Threat Information
  Arms: PMT Threat Appraisal
Behavioral: General Nutrition and Lifestyle — The first half of the PMT absent video will be presented by the Alliance for Aging Research, including an immersive video design, explaining the impact that nutrition may have as the participants age, reviewed by Dr. Steven Austad and Senior Nutritionist Johanna Dwyer. The second half of the PMT absent video will be presented by TED-Ed with narration by Addison Anderson, including a similar immersive video design, explaining how the food the participants eat may affect our brain and overall health. The nutrition and lifestyle information design will be administered as a control because it provides informative lifestyle choices regarding nutrition that can help promote the participants overall health without having an underlying link to vaping behaviour and its subsequent effect on the status of health.
  Other Names: Attention Control; Nutrition and Lifestyle
  Arms: Nutrition and Lifestyle Control

SUMMARY:
Participants will be allocated to one of two experimental groups using a blocked randomization method; participants will be randomized within blocks such that an equal number are assigned to each treatment. Allocation proceeds by randomly selecting one of the orderings and assigning the next block of participants to study groups according to the specific sequence. Once participants are allocated to one block, each block will be randomly assigned to one of the two interventions. Participants will be randomly divided into one of two blocks, each containing a maximum of 75 participants. Possible treatment allocations within each block are (1) AABB, (2) BBAA, (3) ABAB, etc. This method ensures equal treatment allocation within each block. Each participant will then be assigned a number that will represent the participants' block as well as the participants' individual participant ID number (i.e., Participant '100-123' would be in the same group as participant '100-124'). Groups will be assigned using an Excel file to input participants into subsequent groupings and keep track of questionnaire submissions. At baseline, purpose-questionnaires will be distributed to both groups to assess history and experience with vaping and measure intention to vape less along with the "baseline self-reported questionnaires" that will be administered on Day 1 to all participants. At Day 7 (T1), respective participants will be emailed the attached video link and questionnaires and be instructed to complete the surveys after watching the participants' respective videos. The study intervention will be a single site trial delivered as a video link to the email provided by the participant; both intervention videos will play on YouTube and participants will be instructed to complete the surveys immediately after watching the video attached to the email sent to the participants. The participants will complete self-reported questionnaires at 3 follow-up periods after baseline in the 6-week protocol (all questionnaires will be sent by the student investigator (SI) to the email provided by the participants). Self-reported vaping behaviour questionnaires will be managed at baseline, Day 7 (T1), Day 30 (T2), and Day 45 (T3).

DETAILED DESCRIPTION:
Participants will be allocated to one of two experimental groups using a blocked randomization method; participants will be randomized within blocks such that an equal number are assigned to each treatment. Allocation proceeds by randomly selecting one of the orderings and assigning the next block of participants to study groups according to the specific sequence. Once participants are allocated to one block, each block will be randomly assigned to one of the two interventions. Participants will be randomly divided into one of two blocks (A or B), each containing a maximum of 75 participants. Possible treatment allocations within each block are (1) AABB, (2) BBAA, (3) ABAB, etc. This method ensures equal treatment allocation within each block. Each participant will then be assigned an ID number that will represent the participants' block as well as the participants' individual participant ID number (i.e., Participant '100-123' would be in the same group as participant '100-124'). Participants will be provided the participants' ID number via email by the SI when the LOI/C is signed by the study team and sent back to the participant. Groups will be randomly allocated to an intervention group and an Excel file will be used to organize participants into subsequent groupings and keep track of questionnaire submissions. Since the total number of participants is 150, the investigators chose the block randomization method to assign groups equally because it is short enough to prevent imbalance and long enough to prevent guessing allocation in trials. Within the study timeline, the investigators plan to implement the block randomization schema following pre-screening and informed consent processing. To avoid the presence of stratification errors the investigators further plan to review the allocation design before administering study intervention and purpose-questionnaires to prevent participant mismanagement during the protocol. At baseline, purpose-questionnaires will be distributed to both groups to assess the participants' history and experience with vaping and measure the participants' intention to vape less along with the "baseline self-reported questionnaires" that will be administered on Day 1 to all participants. At Day 7 (T1), respective participants will be emailed an attached video link and the questionnaires and be instructed to complete the surveys immediately after watching the video. The study intervention will be a single site trial delivered as a video link to the email provided by the participant; both intervention videos will play on YouTube. The participants will complete self-reported questionnaires at 3 follow-up periods after baseline in the 6-week protocol (all questionnaires will be sent by the student investigator (SI) to the email provided by the participants). Self-reported vaping behaviour questionnaires will be managed at baseline, Day 7 (T1), Day 30 (T2), and Day 45 (T3). All interventions will be created using the Qualtrics Survey Software and will be distributed to the email provided by the individual participants.

The Protection motivation theory is a theory that helps to clarify fear appeals. The protection motivation theory proposes that the participants choose to commit to certain behaviours for self-protection based on four factors: the perceived severity of a threatening event, the perceived probability of the occurrence, or vulnerability, the efficacy of the recommended preventive behaviour, and the perceived self-efficacy. Within the study design, participant groups are one of two treatment conditions: PMT present or PMT absent (attention control). The PMT present group will include an 8-minute informational video that explains the current research and health risks associated with vaping, within the context of a threat appraisal focus (Perceived Vulnerability and Perceived Severity). During this video intervention, the severity of vaping among young adult populations, incorporating both the short and long-term health effects will be presented. In addition, the negative impact of vaping and the lack of research and information that currently exists on popular vaping products will be brought to light, including the potentially devastating impact it can have on the health of young adults. The PMT absent group will feature an 8-minute nutrition and lifestyle information video as an attention control strategy in this study. During this video intervention, the general risks and benefits of nutrition and lifestyle choices will be presented. The focus of this video will be on how a balanced diet and proper lifestyle choices (i.e., adequate sleep) can benefit the participants lives in the short-term and long-term. In regard to lifestyle choices, the topic of substance abuse will be discussed briefly but without depth or research. The reason for the nutrition and lifestyle information group control intervention is because it provides informative lifestyle choices that can help promote the participants overall health without having an underlying link to vaping behaviour, separating and illustrating the impact of the specific information provided by the threat appraisal PMT, compared to general nutrition and lifestyle advice on overall vaping intention and behaviour of a Canadian student population of mostly young adults. Within the study procedures, the investigators acknowledge the potential impact retrospective questionnaires may have on participants; in the study design the investigators expect there to be a change in intention to vape as a result of the intervention, specifically in the PMT group, however, the investigators do not expect the questionnaires alone to cause statistically significant change to participant behaviour-intention or action-behaviour.

If the Principal Investigator (PI) and Student Investigator (SI) determine safe behaviour is not being practiced and/or the participant is not in a stable psychological state, the SI will email the respective participant(s) privately and explain that the participants should only continue to participate in this study if the participants feel safe and psychologically sound. The contact information of a clinical psychologist, Dr. Lisa Lee, and the Counselling Service of London, specialized in anxiety therapy and self-esteem counselling, both as part of the study team, will be included in this email or provided to participants upon request, along with the Center for Addiction and Mental Health (CAMH) distress phone number. The role of Dr. Lee and the Counselling Service of London are to work as a mental health resource for participants in cases that the PI and SI deem the participant is not practicing safe behaviour/in a stable psychological state and in circumstances where the participant requests additional aid from the study team. All participants will also be reminded to contact the participants' respective university health centre resources. In extreme cases, if the SI and PI recognize a participant is continuing to not practice safe behaviour or maintain a stable psychological state, the participant will be withdrawn from study participation and the contact information for Dr. Lee, the Counselling Services of London, and the CAMH distress line will be provided to the participant again, advising the participants to call, email, or text the health and wellness centre for additional aid.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Ability to read and understand English
3. Stated willingness to comply with all study procedures and availability for the duration of the study
4. Males and females; Age 18 years and older
5. Self-report as current users of vaping products (>3x in the past 30 days)
6. Willingness to adhere to the study intervention regimen
7. Enrolled full-time within a registered Canadian university during the 2020-2021 school year
8. Access to necessary resources for participating in a technology-based intervention (i.e., computer, smartphone, internet access)
9. Willingness to stop (or at least decrease the frequency of) vaping

Exclusion Criteria:

1. Activity restrictions that limit one's ability to engage in questionnaire testing
2. Currently practicing in behaviour therapy treatment specific to vaping or attending a rehab centre
3. At the time of signing/submitting this consent form the participants are under the legal age of 18
4. Failure to complete and submit completed questionnaires within the 7-day study timeframe, starting the day that set of surveys is emailed to the participants by the student investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Effect of Threat Appraisal on Vaping Intention | 6-weeks
  Vaping intention was measured at each time-point (baseline (Day 0), T1 (Day 7), T2 (Day 30), T3 (Day 45)) using the threat appraisal Protection Motivation Theory (PMT) questionnaire to assess individuals' relative and immediate feelings about vaping before and after intervention over the 6-week follow-up periods, reporting a score on a scale between 1 and 10, 1 representing a low perceived threat outcome and 10 illustrating a high perceived threat outcome. Threat appraisals within PMT also identified Perceived Vulnerability (PV) and Perceived Severity (PS) of individual participants at each phase of the study protocol in order to assess delayed and processed fear associated with vaping devices, following the intervention. The primary hypothesis is those exposed to the threat appraisal information grounded in the PMT components of severity and vulnerability will score higher on purpose-built questions reflecting these components than their attentional information control counterparts.

SECONDARY OUTCOMES:
Effect of Perceived Vulnerability on Intention | 6-weeks
  Reduction in intentions to vape were dependent on the extent to which individual participants experienced the intervention information. Perceived Vulnerability (PV) questions identified in the Protection Motivation Theory (PMT) questionnaire include items that question the individual participants' experience of their respective videos. Reporting was scored on a scale between 1 and 10, 1 representing a low intention and 10 a high intention to reduce vaping. These appreciations will indicate the power between inter-correlated vulnerability and severity, separately. Greater significance in vaping intention will be cross-examined to determine the influence of PV, independently. The secondary hypothesis is that those exposed to the threat appraisal information grounded in the PMT components of severity and vulnerability will show lower intentions to vape and lower vaping use compared to their attentional information (nutrition and lifestyle information group) control counterpart.
Effect of Perceived Severity on Intention | 6-weeks
  Reduction in intentions to vape were dependent on the extent to which participants experienced the intervention information. Perceived Severity (PS) questions identified in the Protection Motivation Theory (PMT) questionnaire included items that questioned the participants' experiences of their respective videos. Reporting was scored on a scale between 1 and 10, 1 representing a low intention and 10 a high intention to reduce vaping. These appreciations will indicate the power between inter-correlated vulnerability and severity, separately. Greater vaping intention will be cross-examined to determine the influence of PS, independently. In conjunction with perceived vulnerability, the secondary hypothesis is that those exposed to the threat appraisal information grounded in the PMT components of severity and vulnerability will show lower intentions to vape and lower vaping use compared to their attentional information (nutrition and lifestyle information group) control counterpart.

OTHER OUTCOMES:
Effect of intention on Behaviour Outcome | 6-weeks
  Participant vaping behaviour was assessed at each timepoint (Day 0), T1 (Day 7), T2 (Day 30), T3 (Day 45)) using the Youth Vaping Questionnaire (YVQ) to assess how changes in intention to vape less translated to subsequent vaping behaviour patterns. The corroboration between intentions to vape less and reduced vaping behaviours were measured using one, five-point item, at each time-point during the six-week timeframe. Reporting was scored on a scale between 1 and 5,1 representing a low behaviour rate and 5 illustrating a high behaviour rate. The tertiary hypothesis is that reduction in intentions to vape will be associated with lower vaping use.

CONTACTS AND LOCATIONS:
Overall Officials: Harry Prapavessi, Ph.D, Principal Investigator — Professor
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Identifiable data will only be stored on the Personal Vault OneDrive data storage, using BitLocker-encryption for security. Because the research team is using an electronic safety/security system for data storage, following the 7 year retainment period, data will be destroyed by selecting the folders with any identifiable material and deleting them. Next, the student investigator will permanently delete the folders from the recycle bin of the OneDrive system to remove any opportunity of data retrieval.

REFERENCES:
- [Background] Azagba S. E-cigarette use, dual use of e-cigarettes and tobacco cigarettes, and frequency of cannabis use among high school students. Addict Behav. 2018 Apr;79:166-170. doi: 10.1016/j.addbeh.2017.12.028. Epub 2017 Dec 23. PMID 29291507
- [Background] Bein K, Leikauf GD. Acrolein - a pulmonary hazard. Mol Nutr Food Res. 2011 Sep;55(9):1342-60. doi: 10.1002/mnfr.201100279. PMID 21994168
- [Background] Bell K, Keane H. Nicotine control: E-cigarettes, smoking and addiction. Int J Drug Policy. 2012 May;23(3):242-7. doi: 10.1016/j.drugpo.2012.01.006. Epub 2012 Feb 23. PMID 22365155
- [Background] Besaratinia A, Tommasi S. Vaping: A growing global health concern. EClinicalMedicine. 2019 Nov 16;17:100208. doi: 10.1016/j.eclinm.2019.10.019. eCollection 2019 Dec. No abstract available. PMID 31891141
- [Background] Boakye E, Obisesan OH, Osei AD, Dzaye O, Uddin SMI, Hirsch GA, Blaha MJ. The Promise and Peril of Vaping. Curr Cardiol Rep. 2020 Oct 9;22(12):155. doi: 10.1007/s11886-020-01414-x. PMID 33037523
- [Background] Callahan-Lyon P. Electronic cigarettes: human health effects. Tob Control. 2014 May;23 Suppl 2(Suppl 2):ii36-40. doi: 10.1136/tobaccocontrol-2013-051470. PMID 24732161
- [Background] Chadi N, Schroeder R, Jensen JW, Levy S. Association Between Electronic Cigarette Use and Marijuana Use Among Adolescents and Young Adults: A Systematic Review and Meta-analysis. JAMA Pediatr. 2019 Oct 1;173(10):e192574. doi: 10.1001/jamapediatrics.2019.2574. Epub 2019 Oct 7. PMID 31403684
- [Background] Cole AG, Aleyan S, Battista K, Leatherdale ST. Correction to: Trends in youth e-cigarette and cigarette use between 2013 and 2019: insights from repeat cross-sectional data from the COMPASS study. Can J Public Health. 2021 Feb;112(1):70. doi: 10.17269/s41997-020-00441-z. No abstract available. PMID 33174129
- [Background] Czoli CD, Hammond D, White CM. Electronic cigarettes in Canada: prevalence of use and perceptions among youth and young adults. Can J Public Health. 2014 Feb 3;105(2):e97-e102. doi: 10.17269/cjph.105.4119. PMID 24886856
- [Background] Darabseh MZ, Selfe J, Morse CI, Degens H. Is vaping better than smoking for cardiorespiratory and muscle function? Multidiscip Respir Med. 2020 Jul 3;15(1):674. doi: 10.4081/mrm.2020.674. eCollection 2020 Jan 28. PMID 32670575
- [Background] Droulers O, Gallopel-Morvan K, Lacoste-Badie S, Lajante M. The influence of threatening visual warnings on tobacco packaging: Measuring the impact of threat level, image size, and type of pack through psychophysiological and self-report methods. PLoS One. 2017 Sep 14;12(9):e0184415. doi: 10.1371/journal.pone.0184415. eCollection 2017. PMID 28910317
- [Background] Fataar F, Hammond D. The Prevalence of Vaping and Smoking as Modes of Delivery for Nicotine and Cannabis among Youth in Canada, England and the United States. Int J Environ Res Public Health. 2019 Oct 25;16(21):4111. doi: 10.3390/ijerph16214111. PMID 31731420
- [Background] Gaston A, Prapavessis H. Using a combined protection motivation theory and health action process approach intervention to promote exercise during pregnancy. J Behav Med. 2014 Apr;37(2):173-84. doi: 10.1007/s10865-012-9477-2. Epub 2012 Nov 23. PMID 23180287
- [Background] Gay B, Field Z, Patel S, Alvarez RM, Nasser W, Madruga M, Carlan SJ. Vaping-Induced Lung Injury: A Case of Lipoid Pneumonia Associated with E-Cigarettes Containing Cannabis. Case Rep Pulmonol. 2020 Apr 3;2020:7151834. doi: 10.1155/2020/7151834. eCollection 2020. PMID 32309002
- [Background] Giovino GA, Mirza SA, Samet JM, Gupta PC, Jarvis MJ, Bhala N, Peto R, Zatonski W, Hsia J, Morton J, Palipudi KM, Asma S; GATS Collaborative Group. Tobacco use in 3 billion individuals from 16 countries: an analysis of nationally representative cross-sectional household surveys. Lancet. 2012 Aug 18;380(9842):668-79. doi: 10.1016/S0140-6736(12)61085-X. PMID 22901888
- [Background] Goniewicz ML, Knysak J, Gawron M, Kosmider L, Sobczak A, Kurek J, Prokopowicz A, Jablonska-Czapla M, Rosik-Dulewska C, Havel C, Jacob P 3rd, Benowitz N. Levels of selected carcinogens and toxicants in vapour from electronic cigarettes. Tob Control. 2014 Mar;23(2):133-9. doi: 10.1136/tobaccocontrol-2012-050859. Epub 2013 Mar 6. PMID 23467656
- [Background] Gravely S, Driezen P, Ouimet J, Quah ACK, Cummings KM, Thompson ME, Boudreau C, Hammond D, McNeill A, Borland R, Thrasher JF, Edwards R, Omar M, Hitchman SC, Yong HH, Barrientos-Gutierrez T, Willemsen MC, Bianco E, Boado M, Goma FM, Seo HG, Nargis N, Jiang Y, Perez CA, Fong GT. Prevalence of awareness, ever-use and current use of nicotine vaping products (NVPs) among adult current smokers and ex-smokers in 14 countries with differing regulations on sales and marketing of NVPs: cross-sectional findings from the ITC Project. Addiction. 2019 Jun;114(6):1060-1073. doi: 10.1111/add.14558. Epub 2019 Feb 20. PMID 30681215
- [Background] Hajek P, Phillips-Waller A, Przulj D, Pesola F, Myers Smith K, Bisal N, Li J, Parrott S, Sasieni P, Dawkins L, Ross L, Goniewicz M, Wu Q, McRobbie HJ. A Randomized Trial of E-Cigarettes versus Nicotine-Replacement Therapy. N Engl J Med. 2019 Feb 14;380(7):629-637. doi: 10.1056/NEJMoa1808779. Epub 2019 Jan 30. PMID 30699054
- [Background] Hammond D, Reid JL, Rynard VL, Fong GT, Cummings KM, McNeill A, Hitchman S, Thrasher JF, Goniewicz ML, Bansal-Travers M, O'Connor R, Levy D, Borland R, White CM. Prevalence of vaping and smoking among adolescents in Canada, England, and the United States: repeat national cross sectional surveys. BMJ. 2019 Jun 20;365:l2219. doi: 10.1136/bmj.l2219. PMID 31221636
- [Background] Jackson CD, Carter J, Kansagara D. E-Cigarettes Versus Nicotine Replacement Therapy for Smoking Cessation : Hajek P, Phillips-waller A, Przulj D, et al. A Randomized Trial of E-Cigarettes versus Nicotine-Replacement Therapy. N Engl J Med. 2019;380(7):629-637. J Gen Intern Med. 2021 May;36(5):1481-1483. doi: 10.1007/s11606-020-06408-7. Epub 2021 Feb 9. No abstract available. PMID 33564946
- [Background] Jakobsen JC, Gluud C, Wetterslev J, Winkel P. When and how should multiple imputation be used for handling missing data in randomised clinical trials - a practical guide with flowcharts. BMC Med Res Methodol. 2017 Dec 6;17(1):162. doi: 10.1186/s12874-017-0442-1. PMID 29207961
- [Background] Jones CL, Jensen JD, Scherr CL, Brown NR, Christy K, Weaver J. The Health Belief Model as an explanatory framework in communication research: exploring parallel, serial, and moderated mediation. Health Commun. 2015;30(6):566-76. doi: 10.1080/10410236.2013.873363. Epub 2014 Jul 10. PMID 25010519
- [Background] Kasza KA, Ambrose BK, Conway KP, Borek N, Taylor K, Goniewicz ML, Cummings KM, Sharma E, Pearson JL, Green VR, Kaufman AR, Bansal-Travers M, Travers MJ, Kwan J, Tworek C, Cheng YC, Yang L, Pharris-Ciurej N, van Bemmel DM, Backinger CL, Compton WM, Hyland AJ. Tobacco-Product Use by Adults and Youths in the United States in 2013 and 2014. N Engl J Med. 2017 Jan 26;376(4):342-353. doi: 10.1056/NEJMsa1607538. PMID 28121512
- [Background] Macdonell K, Chen X, Yan Y, Li F, Gong J, Sun H, Li X, Stanton B. A Protection Motivation Theory-Based Scale for Tobacco Research among Chinese Youth. J Addict Res Ther. 2013 Jul 8;4:154. doi: 10.4172/2155-6105.1000154. PMID 24478933
- [Background] Maclaren DJ, Conigrave KM, Robertson JA, Ivers RG, Eades S, Clough AR. Using breath carbon monoxide to validate self-reported tobacco smoking in remote Australian Indigenous communities. Popul Health Metr. 2010 Feb 20;8(1):2. doi: 10.1186/1478-7954-8-2. PMID 20170528
- [Background] Masiero M, Cutica I, Russo S, Mazzocco K, Pravettoni G. Psycho-cognitive predictors of burnout in healthcare professionals working in emergency departments. J Clin Nurs. 2018 Jul;27(13-14):2691-2698. doi: 10.1111/jocn.14376. Epub 2018 Jun 1. PMID 29856096
- [Background] McRobbie H. Modelling the Population Health Effects of E-Cigarettes Use: Current Data Can Help Guide Future Policy Decisions. Nicotine Tob Res. 2017 Feb;19(2):131-132. doi: 10.1093/ntr/ntw387. Epub 2016 Dec 24. No abstract available. PMID 28013269
- [Background] The Lancet Respiratory Medicine. The EVALI outbreak and vaping in the COVID-19 era. Lancet Respir Med. 2020 Sep;8(9):831. doi: 10.1016/S2213-2600(20)30360-X. Epub 2020 Aug 14. No abstract available. PMID 32805203
- [Background] Morello P, Perez A, Pena L, Lozano P, Thrasher JF, Sargent JD, Mejia R. PREVALENCE AND PREDICTORS OF E-CIGARETTE TRIAL AMONG ADOLESCENTS IN ARGENTINA. Tob Prev Cessat. 2016 Dec;2:80. doi: 10.18332/tpc/66950. PMID 31355353
- [Background] Ogunwale MA, Li M, Ramakrishnam Raju MV, Chen Y, Nantz MH, Conklin DJ, Fu XA. Aldehyde Detection in Electronic Cigarette Aerosols. ACS Omega. 2017 Mar 31;2(3):1207-1214. doi: 10.1021/acsomega.6b00489. Epub 2017 Mar 29. PMID 28393137
- [Background] Olmedo P, Goessler W, Tanda S, Grau-Perez M, Jarmul S, Aherrera A, Chen R, Hilpert M, Cohen JE, Navas-Acien A, Rule AM. Metal Concentrations in e-Cigarette Liquid and Aerosol Samples: The Contribution of Metallic Coils. Environ Health Perspect. 2018 Feb 21;126(2):027010. doi: 10.1289/EHP2175. PMID 29467105
- [Background] Pechacek TF, Nayak P, Gregory KR, Weaver SR, Eriksen MP. The Potential That Electronic Nicotine Delivery Systems Can be a Disruptive Technology: Results From a National Survey. Nicotine Tob Res. 2016 Oct;18(10):1989-1997. doi: 10.1093/ntr/ntw102. Epub 2016 May 3. PMID 27142201
- [Background] Peruzzi M, Biondi-Zoccai G, Carnevale R, Cavarretta E, Frati G, Versaci F. Vaping Cardiovascular Health Risks: an Updated Umbrella Review. Curr Emerg Hosp Med Rep. 2020;8(3):103-109. doi: 10.1007/s40138-020-00219-0. Epub 2020 Jun 16. PMID 32837803
- [Background] Prapavessis H, De Jesus S, Fitzgeorge L, Faulkner G, Maddison R, Batten S. Exercise to Enhance Smoking Cessation: the Getting Physical on Cigarette Randomized Control Trial. Ann Behav Med. 2016 Jun;50(3):358-69. doi: 10.1007/s12160-015-9761-9. PMID 26791022
- [Background] Rogers RW. A Protection Motivation Theory of Fear Appeals and Attitude Change1. J Psychol. 1975 Sep;91(1):93-114. doi: 10.1080/00223980.1975.9915803. PMID 28136248
- [Background] Ruiter RA, Kok G, Verplanken B, Brug J. Evoked fear and effects of appeals on attitudes to performing breast self-examination: an information-processing perspective. Health Educ Res. 2001 Jun;16(3):307-19. doi: 10.1093/her/16.3.307. PMID 11497114
- [Background] Sadeghi R, Mazloomy Mahmoodabad SS, Fallahzadeh H, Rezaeian M, Bidaki R, Khanjani N. Hookah is the enemy of health campaign: a campaign for prevention of hookah smoking among youth. Health Promot Int. 2020 Oct 1;35(5):1125-1136. doi: 10.1093/heapro/daz109. PMID 31687738
- [Background] Sassano MF, Davis ES, Keating JE, Zorn BT, Kochar TK, Wolfgang MC, Glish GL, Tarran R. Evaluation of e-liquid toxicity using an open-source high-throughput screening assay. PLoS Biol. 2018 Mar 27;16(3):e2003904. doi: 10.1371/journal.pbio.2003904. eCollection 2018 Mar. PMID 29584716
- [Background] Sheeran P, Orbell S. Using implementation intentions to increase attendance for cervical cancer screening. Health Psychol. 2000 May;19(3):283-9. doi: 10.1037//0278-6133.19.3.283. PMID 10868773
- [Background] Siegel MB, Tanwar KL, Wood KS. Electronic cigarettes as a smoking-cessation: tool results from an online survey. Am J Prev Med. 2011 Apr;40(4):472-5. doi: 10.1016/j.amepre.2010.12.006. PMID 21406283
- [Background] Silagy C, Mant D, Fowler G, Lodge M. Meta-analysis on efficacy of nicotine replacement therapies in smoking cessation. Lancet. 1994 Jan 15;343(8890):139-42. doi: 10.1016/s0140-6736(94)90933-4. PMID 7904003
- [Background] Silver B, Ripley-Moffitt C, Greyber J, Goldstein AO. Successful use of nicotine replacement therapy to quit e-cigarettes: lack of treatment protocol highlights need for guidelines. Clin Case Rep. 2016 Mar 11;4(4):409-11. doi: 10.1002/ccr3.477. eCollection 2016 Apr. PMID 27099740
- [Background] Teasdale JE, Newby AC, Timpson NJ, Munafo MR, White SJ. Cigarette smoke but not electronic cigarette aerosol activates a stress response in human coronary artery endothelial cells in culture. Drug Alcohol Depend. 2016 Jun 1;163:256-60. doi: 10.1016/j.drugalcdep.2016.04.020. Epub 2016 Apr 22. PMID 27137404
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Thrul J, Stemmler M, Buhler A, Kuntsche E. Adolescents' protection motivation and smoking behaviour. Health Educ Res. 2013 Aug;28(4):683-91. doi: 10.1093/her/cyt062. Epub 2013 Jun 13. PMID 23766453
- [Background] Tommasi S, Caliri AW, Caceres A, Moreno DE, Li M, Chen Y, Siegmund KD, Besaratinia A. Deregulation of Biologically Significant Genes and Associated Molecular Pathways in the Oral Epithelium of Electronic Cigarette Users. Int J Mol Sci. 2019 Feb 10;20(3):738. doi: 10.3390/ijms20030738. PMID 30744164
- [Background] Trtchounian A, Williams M, Talbot P. Conventional and electronic cigarettes (e-cigarettes) have different smoking characteristics. Nicotine Tob Res. 2010 Sep;12(9):905-12. doi: 10.1093/ntr/ntq114. Epub 2010 Jul 19. PMID 20644205
- [Background] Tulloch H, Reida R, D'Angeloa MS, Plotnikoff RC, Morrina L, Beatona L, Papadakisa S, Pipe A. Predicting short and long-term exercise intentions and behaviour in patients with coronary artery disease: A test of protection motivation theory. Psychol Health. 2009 Mar;24(3):255-69. doi: 10.1080/08870440701805390. PMID 20204992
- [Background] National Center for Chronic Disease Prevention and Health Promotion (US) Office on Smoking and Health. E-Cigarette Use Among Youth and Young Adults: A Report of the Surgeon General [Internet]. Atlanta (GA): Centers for Disease Control and Prevention (US); 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK538680/ PMID 30869850
- [Background] van de Ven K, Ritter A, Berends L, Chalmers J, Lancaster K. Perceptions of purchasing and payment mechanisms in alcohol and other drug treatment services in Australia: A qualitative study involving alcohol and other drug service providers and purchasers of treatment. Drug Alcohol Rev. 2020 Feb;39(2):189-197. doi: 10.1111/dar.13027. PMID 32012374
- [Background] Weinstein ND. The precaution adoption process. Health Psychol. 1988;7(4):355-86. doi: 10.1037//0278-6133.7.4.355. PMID 3049068
- [Background] Iacobucci G. WHO calls for ban on e-cigarette use indoors. BMJ. 2014 Aug 27;349:g5335. doi: 10.1136/bmj.g5335. No abstract available. PMID 25170124
- [Background] Worsley DJ, Jones K, Marshman Z. Patients are asking about e-cigarettes. What do we tell them? Br Dent J. 2014 Jul;217(2):91-5. doi: 10.1038/sj.bdj.2014.596. PMID 25060461
- [Background] Wu CS, Wong HT, Chou LY, To BP, Lee WL, Loke AY. Correlates of Protective Motivation Theory (PMT) to adolescents' drug use intention. Int J Environ Res Public Health. 2014 Jan 3;11(1):671-84. doi: 10.3390/ijerph110100671. PMID 24394215
- [Background] Xie W, Kathuria H, Galiatsatos P, Blaha MJ, Hamburg NM, Robertson RM, Bhatnagar A, Benjamin EJ, Stokes AC. Association of Electronic Cigarette Use With Incident Respiratory Conditions Among US Adults From 2013 to 2018. JAMA Netw Open. 2020 Nov 2;3(11):e2020816. doi: 10.1001/jamanetworkopen.2020.20816. PMID 33180127
- [Background] Yan Y, Jacques-Tiura AJ, Chen X, Xie N, Chen J, Yang N, Gong J, Macdonell KK. Application of the protection motivation theory in predicting cigarette smoking among adolescents in China. Addict Behav. 2014 Jan;39(1):181-8. doi: 10.1016/j.addbeh.2013.09.027. Epub 2013 Oct 2. PMID 24157424
- [Background] Zhao Z, Zhang M, Wu J, Xu X, Yin P, Huang Z, Zhang X, Zhou Y, Zhang X, Li C, Wang L, Gao GF, Wang L, Li X, Zhou M. E-cigarette use among adults in China: findings from repeated cross-sectional surveys in 2015-16 and 2018-19. Lancet Public Health. 2020 Dec;5(12):e639-e649. doi: 10.1016/S2468-2667(20)30145-6. PMID 33271077
- See also: Growth in Popularity of Vaping — https://time.com/3590093/oxfords-2014-word-of-the-year-is-vape/
- See also: Trend of Vaping in North America — https://www.grandviewresearch.com/industry-analysis/us-e-cigarette-vape-market
- See also: International Vaping Statistics — https://www.statista.com/statistics/978458/users-electronic-cigarette-france/

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT04982978/Prot_SAP_ICF_000.pdf